CLINICAL TRIAL: NCT03652558
Title: The Effects of Ozone Therapy as an Adjunct to Periodontal Treatment: A Randomized Split-Mouth Clinical Trial
Brief Title: Effects of Ozone Therapy as an Adjunct to Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zekeriya Tasdemir, Principal investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tasdemir
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: In this study the investigators select the split mouth study design to eleminate host effects on healing.
Who Masked: Participant, Investigator
Masking Description: Investigators who evaluate the clinical and biochemical parameters did no know the groups.
  And participants did not know ozone device work or not when holding the probe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone group (Experimental): topical gaseous ozone was applied into periodontal pockets during active periodontal therapy
  Interventions: Device: Ozone application with the Ozonytron XL device
- non-ozone group (No Intervention): Only active periodontal therapy was performed

INTERVENTIONS:
Device: Ozone application with the Ozonytron XL device — An ozone generator (Ozonytron; Bionix, Munchen, Germany) with an KPX probe (CA Probe; Ozonytron, Bionix, Munchen, Germany) was used for OT. Topical gaseous ozone was applied into the periodontal pocket twice a week for 2 weeks based on the manufacturer's instructions. Ozone applications were at 75% power for 30 seconds (75 µg/ml). Ozone applications were performed by an experienced investigator. Ozone applications in the control side were simulated without starting the ozone generator
  Arms: ozone group

SUMMARY:
This randomized, placebo controlled, split-mouth clinical study trial evaluates the effects of Ozone therapy on clinical and biochemical parameters. Total of 20 participants completed the study . Periodontal parameters were evaluated at baseline and 3 months following periodontal therapy. All participants were treated non-surgically. Topical gaseous ozone was applied into periodontal pockets. Gingival crevicular fluid pentraxin-3 (PTX-3), interleukin-1β (IL-1β) and high sensitivity C-reactive protein (Hs-CRP) were evaluated.

DETAILED DESCRIPTION:
Ozone therapy (OT) is very popular in medicine. Especially it use for wound healing and antibacterial properties. This randomized, placebo controlled, randomized split-mouth clinical study evaluates the effects of ozone therapy on clinical and biochemical parameters. Total of 20 participants completed the study (10 males, 10 females). Periodontal parameters, including plaque index (PI), gingival index (GI), probing depth (PD), percentage of bleeding on probing, percentage of pockets deeper than 5 mm and clinical attachment level (CAL), and percentage of ≥3 mm clinical attachment level. Periodontal parameters were evaluated at baseline and 3 months following periodontal therapy. All participants were treated non-surgically. Topical gaseous ozone was applied into periodontal pockets twice a week for 2 weeks during active periodontal therapy. Gingival crevicular fluid pentraxin-3 (PTX-3), interleukin-1β (IL-1β) and high sensitivity C-reactive protein (Hs-CRP) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years of age
* Generalized chronic periodontitis(Armitage, 1999)
* Systemically healthy
* More than 20 teeth (excluding third molars)

Exclusion Criteria:

* Periodontal treatment within 6 months
* Antibiotic use within the previous 3 months
* Pregnancy and lactation
* Past or current smoking and alcohol consumption
* Contraindications for OT
* Patients with class II and III furcation defects(Staffileno, 1969)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Periodontal disease parameters change | Examinations were performed at baseline and 3 months after periodontal therapy. Changes is determined with baseline values - 3 months after periodontal treatment.
  Probing depth (mm) were evaluated by periodontal probe.

SECONDARY OUTCOMES:
Gingival crevicular inflammatory parameter change | inflammatory biochemical parameters were analyzed at baseline and 3 months after periodontal therapy and changes is determined with baseline values - 3 months after periodontal therapy.
  Gingival crevicular fluid pentraxin-3 (PTX-3) ng/mL was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Zekeriya Taşdemir, Phd, Principal Investigator — TC Erciyes University

IPD SHARING:
Plan to Share IPD: Undecided